CLINICAL TRIAL: NCT03177668
Title: Phase I/II Clinical Study of YS110 in Patients With Malignant Pleural Mesothelioma
Brief Title: Clinical Study of YS110 in Patients With Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YS1101
Record Dates: First submitted 2017-05-23; First posted 2017-06-06 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YS110 (Experimental): Phase 1 part: Administration of 3 different dose cohort
  Phase 2 part: Administration of recommended dose determined from result of Phase 1 part
  Interventions: Drug: YS110

INTERVENTIONS:
Drug: YS110 — Intravenous administration

SUMMARY:
The purpose of this study is to examine tolerability, safety, and pharmacokinetics of YS110 intravenous administration in patients with malignant pleural mesothelioma and to preliminarily examine the anti-tumor effect of YS110.

ELIGIBILITY:
Inclusion Criteria:

* Patient with male or female aged ≥ 20 (and aged < 75 in Phase 1 part)
* Patients whose malignant pleural mesothelioma was histologically confirmed
* Patients who have advanced pleural mesothelioma that are refractory to existing anti-tumor drugs and who have no other standard therapies which should be prioritized
* Patients whose most recent major surgery (except exploratory thoracotomy or laparotomy) or drug or radiation therapy for malignant tumors, if any, was at least 4 weeks ago (at least 12 weeks ago for immunotherapy) at the subject enrollment
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 1 or less

Exclusion Criteria:

* Patients whose toxicity findings in the previous treatment (antineoplastic agents) have not been yet restored
* Patients with tumor lesions in central nervous system confirmed in MRI or CT

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Status of onset of Dose Limiting Toxicity (DLT) | 18 days
  Assessed by number of subjects with DLT of YS110
Disease Control Rate (DCR) | 6 months
  The proportion of subjects with assessed overall response as Complete Response (CR), Partial Response (PR) or Stable Disease (SD)
Progression Free Survival (PFS) | Assessed for duration of study participation which is estimated to be 18 months
  The period from the starting day of the administration to Progressive Disease (PD) or death
Response Rate (RR) | Assessed for duration of study participation which is estimated to be 18 months
  The proportion of subjects with assessed the best overall response as CR or PR
Overall Survival (OS) | Assessed for duration of study participation which is estimated to be 18 months
  The period from the starting day of the administration to death
LCSS-Meso | Assessed for duration of study participation which is estimated to be 18 months
  Assessed for Quality of life (QOL) by using the modified Lung Cancer Symptom Scale for mesothelioma
EORTC QLQ-C30 | Assessed for duration of study participation which is estimated to be 18 months
  Assessed for QOL by using the Japanese versions of EORTC QLQ-C30 in the cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Nobuo Kanai, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Research Site, Multiple Locations, Japan